CLINICAL TRIAL: NCT02935309
Title: Phase I Study of Pre-operative Capecitabine and Lenvatinib With External Radiation Therapy in Locally Advanced Rectal Adenocarcinoma
Brief Title: Capecitabine and Lenvatinib With External Radiation in Rectal Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18646
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Rectal Cancer; Rectal Adenocarcinoma
Keywords: rectum; transrectal; carcinoma
MeSH Terms: conditions — Rectal Neoplasms; Carcinoma | interventions — lenvatinib; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pre-Surgery Chemotherapy/Radiotherapy (Experimental): Pre-surgery chemotherapy and external radiation therapy. Dose escalation of Lenvatinib; fixed dose Capecitabine; Radiotherapy. Lenvatinib and capecitabine will be started on day 1 with radiation and will be discontinued on the last day of radiation. Surgical resection should occur between 6 - 10 weeks after the participant completes preoperative lenvatinib, capecitabine, and radiation therapy. Postoperative chemotherapy after surgery will be given at investigator's discretion.
  Interventions: Drug: Lenvatinib; Drug: Capecitabine; Radiation: External Radiation Therapy (XRT)

INTERVENTIONS:
Drug: Lenvatinib — Pre-surgery Lenvatinib, days 1 - 5. Dose Escalation Levels: 1.) 10 mg by mouth (PO) daily (QD); 2.) 14 mg PO QD; 3.) 20 mg PO QD; 4.) 24 PO QD.
  Other Names: E7080
Drug: Capecitabine — Pre-surgery Capecitabine, 850 mg/m^2, twice a day (BID) on days 1-5 for 5½ -6 weeks.
  Other Names: Teva-Capecitabine; Xeloda
Radiation: External Radiation Therapy (XRT) — Pre-surgery RT: Participants will receive 6 weeks of radiation therapy. The radiation sessions will be daily, Monday through Friday, except for holidays.
  Other Names: Radiotherapy; Radiation Therapy (RT)

SUMMARY:
This research study is designed to see if Capecitabine and Lenvatinib in combination with external radiation therapy are effective in treating locally advanced rectal adenocarcinoma in patients who have not yet had surgery, and what the best dosage is.

ELIGIBILITY:
Inclusion Criteria:

* Histologically (archival tissue) confirmed adenocarcinoma of the rectum that begins within 12 cm of the anal verge as determined by sigmoidoscopy and/or colonoscopy with no evidence of distant metastasis.
* Locally advanced rectal cancer determined by any of the following features: 1.) Fixed or immobile tumor on physical exam and/or; 2.) T3 disease with invasion through the muscularis propria as defined by transrectal ultrasound, CT or MRI; 3.) T4 disease with invasion of adjacent structures such as pelvic sidewall, sacrum, pelvis, bladder and/or prostate as determined appropriate imaging modalities such as ultrasound, CT or MRI; 4.) Any T with + N on CT scan/MRI or transrectal ultrasound.
* Age equal to or greater than 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Adequate bone marrow, liver and renal function.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least 3 months after the last administration of lenvatinib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria:

* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Participants must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Previous pelvic irradiation therapy.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
* Active clinically serious infection > CTCAE Grade 2.
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic, attacks, deep vein thrombosis (DVT) within the past 6 months.
* Bleeding or thrombotic disorders or use of anticoagulants, such as warfarin, or similar agents requiring therapeutic international normalized ration (INR) monitoring. (Treatment with low molecular weight heparin (LMWH) is allowed).
* Active malignancy except for non-melanoma skin cancer or in situ cervical cancer or treated non-pelvic cancer from which the patient has been continuously disease free more than 3 years.
* Marked baseline prolongation of QT/QTc interval (QTc interval ≥ 500 msec) using the Fridericia method (QTc = QT/RR0.33) for QTc analysis.
* Greater than 30 mg/dL on urine analysis. Patients with >30 mg/dL on urine analysis on urine analysis will undergo 24-hour urine collection for quantitative assessment of proteinuria. Patients with 24-hour protein ≥1 g/24 hours will be ineligible.
* Needing medical attention for serious bleeding in past 4 weeks.
* Previous chemotherapy except for antiangiogenic agent or tyrosine kinase inhibitor (TKI) will be allowed as long as it is more than 5 years.
* Major surgeries within 3 weeks of starting chemotherapy.
* Evidence or history of bleeding diathesis.
* Use of St. John's Wort or rifampin.
* Known or suspected allergy to lenvatinib or any agent given in the course of this trial.
* Any condition that impairs participant's ability to swallow whole pills.
* Any malabsorption problem.
* Medical need for the continued use of potent inhibitors/inducers of CYP3A4.
* Creatinine clearance not within study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 6 months
  MTD of lenvatinib used in combination with capecitabine and external beam radiation as neoadjuvant therapy for patients with locally advanced rectal carcinoma. The MTD of lenvatinib will be defined as the highest dose level at which no more than 1 out of 6 participants experiences dose-limiting toxicity (DLT). DLT: Any of the hematology or non-hematologic toxicities noted in Table 3 of the protocol, considered to be at least possibly related to lenvatinib and/or capecitabine.

SECONDARY OUTCOMES:
Rate of Pathologic Response | Up to 36 months
  Pathologic response rate after pre-operative therapy and surgery. Pathologic Complete Response (pCR) will be defined as pathologic proof of a complete response based on histologic evaluation of the resected specimen.
Occurrence of Treatment Related Adverse Events | Up to 36 months
  To further define safety profile of the combination. Adverse events will be graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0.

OTHER OUTCOMES:
Rate of Potential Biomarkers for Vascular Endothelial Growth Factor (VEGF) | Up to 36 months
  Investigators will identify potential biomarkers for VEGF pathway and attempt to correlate with pCR. The associations of the potential biomarkers and radiosensitivity index (RSI) with pCR will be examined using logistic regression. A two-sided p-value of <0.05 will be considered statistically significant.
Radiosensitivity Index (RSI) | Up to 36 months
  To determine if low radiosensitivity index (RSI) will correlate with pathologic complete response (pCR). pCR will be examined using logistic regression. A two-sided p-value of <0.05 will be considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Mehta R, Frakes J, Kim J, Nixon A, Liu Y, Howard L, Martinez Jimenez ME, Carballido E, Imanirad I, Sanchez J, Dessureault S, Xie H, Felder S, Sahin I, Hoffe S, Malafa M, Kim R. Phase I Study of Lenvatinib and Capecitabine with External Radiation Therapy in Locally Advanced Rectal Adenocarcinoma. Oncologist. 2022 Aug 5;27(8):621-e617. doi: 10.1093/oncolo/oyac003. PMID 35325225
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/